CLINICAL TRIAL: NCT06413524
Title: The Effects of Different Vibration Exercises on the Strength of Lower Extremity Muscles, Exercise Endurance, and Quality of Life Among COPD Patients
Brief Title: The Effects of Different Vibration Exercises on COPD Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University (Other)
Collaborators: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: N202403010
Record Dates: First submitted 2024-05-09; First posted 2024-05-14 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: COPD; COPD Chronic Obstructive Pulmonary Disease; Vibration Therapy
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

ARMS (3):
- Whole-body Vibration Training Group (Experimental): Receive whole-body vibration twice a week for 12 weeks.
  Interventions: Device: Whole-body Vibration Therapy
- Local Vibration Training Group (Experimental): Receive local vibration twice a week for 12 weeks.
  Interventions: Device: Local Vibration Therapy
- Control Group (No Intervention): Receive no intervention

INTERVENTIONS:
Device: Whole-body Vibration Therapy — Each session includes six series, each lasting 2 minutes, with a frequency of 35 Hz and an amplitude of 2 mm, with a 60-second rest interval between series. For the starting position, the patient stands relaxed on the platform, holding the WBV platform handles.
  Arms: Whole-body Vibration Training Group
Device: Local Vibration Therapy — Each session includes six series, each lasting 2 minutes, with a frequency of 35 Hz and an amplitude of 2 mm, with a 60-second rest interval between series. After the warm-up exercise, the researcher helps the patient wear the localized vibration instrument. During the vibration, participants will hold onto the handle to ensure balance stability.
  Arms: Local Vibration Training Group

SUMMARY:
Pulmonary rehabilitation is effective in improving exercise tolerance, dyspnea, and fatigue in patients with COPD, and exercise training is an important component of pulmonary rehabilitation. Vibration training can be used as a supplement or alternative to traditional exercise and is a short, safe rehabilitation training.

COPD patients will be recruited and randomly assigned to the control group, whole-body vibration training group, or local vibration training group. The study aims to confirm the rehabilitative benefits of enhancing lower limb muscle strength, exercise endurance, and the quality of life related to COPD in patients.

DETAILED DESCRIPTION:
Background Pulmonary rehabilitation is effective in improving exercise tolerance, dyspnea, and fatigue in patients with COPD, and exercise training is an important component of pulmonary rehabilitation. Vibration training can be used as a supplement or alternative to traditional exercise and is a short, safe rehabilitation training.

Purpose To enhance the effectiveness of pulmonary rehabilitation, the vibration rehabilitation system will be applied on COPD patients to validate the effectiveness of direct and indirect vibration interventions on lower extremity muscle strength and functional performance in COPD patients, and test the effectiveness of vibration in improving lower extremity muscle strength, exercise tolerance, and COPD- related quality of life in COPD patients.

Methods COPD patients will be recruited and randomly assigned to the control group, whole-body vibration training group, or local vibration training group. The study aims to confirm the rehabilitative benefits of enhancing lower limb muscle strength, exercise endurance, and the quality of life related to COPD in patients.

Expected outcome To establish an optimal model for lower extremity vibration and to validate the effectiveness of direct vibration on the lower extremities and whole body vibration in COPD patients undergoing pulmonary rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 40.
2. Diagnosis of chronic obstructive pulmonary disease (COPD) based on the criteria established by the Global Initiative for Chronic Obstructive Lung Disease (GOLD).
3. Disease Severity: FEV1 < 50% or COPD patients who have used systemic corticosteroids due to an acute exacerbation of COPD within the past year and are currently in a stable condition.
4. Willingness to participate in vibration exercise intervention and ability to comply with the study activities, including signing the informed consent form.
5. Clear consciousness, normal cognitive function, and ability to communicate in Mandarin or Taiwanese for understanding experimental procedures and relevant instructions.

Exclusion Criteria:

1. Engages in regular physical activity, exercising at least 3 times a week for over 30 minutes, with a Borg Scale rating of 3 for breathlessness after exercise.
2. The interval since the last pulmonary rehabilitation is less than three months.
3. Contraindications to vibration therapy: pregnancy, cardiovascular diseases (with a pacemaker or stent), intervertebral disc diseases, tendinitis, arthritis, hernia, presence of tumors, orthopedic or trauma-related conditions, epilepsy, history of deep vein thrombosis, patients with internal implants.
4. Inability to undergo training or walk due to physical factors, such as being bedridden for an extended period, relying on a ventilator for an extended period, prone to dizziness, central nervous system disorders, etc.
5. Underwent lower limb-related surgery within the past year or is in the recovery period post-surgery.
6. Currently diagnosed with cancer or undergoing cancer treatment.
7. Participation in other research studies.

Ages: 40 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2024-08-08 (Actual); Primary Completion 2025-04-21 (Estimated); Study Completion 2025-06-13 (Estimated)

PRIMARY OUTCOMES:
6 Minute Walking Test | Base line, Week12, Week16
  This test measures how far the patient can walk in 6 minutes, with a greater distance indicating better performance.
Maximal voluntary contraction force | Base line, Week12, Week16
  The readings from the digital dynamometer can be converted into kilograms, with higher values indicating greater muscle strength.

SECONDARY OUTCOMES:
Five Times Sit to Stand Test (FTSST) | Base line, Week12, Week16
  Score is the amount of time it takes for an patient to transfer from a seated position to standing position and back to sitting five times. A shorter time indicates better performance.
Clinical COPD Questionnaire score, CCQ | Base line, Week12, Week16
  The scale ranges from 0 to 6, where higher scores reflect more severe conditions.
  Score Range:
  0: No impact or impairment. 6: Severe impact or impairment.
COPD assessment Test, CAT | Base line, Week12, Week16
  CAT has a scoring range of zero to 40; higher scores indicate a greater severity of COPD's impact on a patient's life.
mMRC dyspnea scale, mMRC | Base line, Week12, Week16
  The scale ranges from 0 to 4, with higher scores representing more severe conditions.

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Medical University WanFang Hospital, Taipei, Wenshan Dist, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] DadeMatthews OO, Agostinelli PJ, Neal FK, Oladipupo SO, Hirschhorn RM, Wilson AE, Sefton JM. Systematic review and meta-analyses on the effects of whole-body vibration on bone health. Complement Ther Med. 2022 May;65:102811. doi: 10.1016/j.ctim.2022.102811. Epub 2022 Jan 29. PMID 35093509
- [Background] Iodice P, Bellomo RG, Gialluca G, Fano G, Saggini R. Acute and cumulative effects of focused high-frequency vibrations on the endocrine system and muscle strength. Eur J Appl Physiol. 2011 Jun;111(6):897-904. doi: 10.1007/s00421-010-1677-2. Epub 2010 Nov 10. PMID 21063726
- [Background] Gupta N, Pinto LM, Morogan A, Bourbeau J. The COPD assessment test: a systematic review. Eur Respir J. 2014 Oct;44(4):873-84. doi: 10.1183/09031936.00025214. Epub 2014 Jul 3. PMID 24993906
- [Background] Djibo DA, Goldstein J, Ford JG. Prevalence of disability among adults with chronic obstructive pulmonary disease, Behavioral Risk Factor Surveillance System 2016-2017. PLoS One. 2020 Feb 27;15(2):e0229404. doi: 10.1371/journal.pone.0229404. eCollection 2020. PMID 32106254
- [Background] Berner K, Albertyn SCS, Dawnarain S, Hendricks LJ, Johnson J, Landman A, Burger M. The effectiveness of combined lower limb strengthening and whole-body vibration, compared to strengthening alone, for improving patient-centred outcomes in adults with COPD: A systematic review. S Afr J Physiother. 2020 Jun 11;76(1):1412. doi: 10.4102/sajp.v76i1.1412. eCollection 2020. PMID 32671277